CLINICAL TRIAL: NCT03238963
Title: A Randomized, Double-masked, Placebo-controlled Exploratory Study to Evaluate Safety, Tolerability, Pharmacodynamics and Pharmacokinetics of Orally Administered BI 1467335 for 12 Weeks With a 12 Week Follow up Period in Patients With Non-proliferative Diabetic Retinopathy Without Center-involved Diabetic Macular Edema (ROBIN Study)
Brief Title: A Study That Tests BI 1467335 in Patients With Diabetic Eye Disease (Diabetic Retinopathy). It Looks at the Way BI 1467335 is Taken up, the Effects it Has, and How Well it is Tolerated.
Acronym: ROBIN
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1386-0012; 2016-002971-91 (EudraCT Number); 1386.12 (Other: Company)
Record Dates: First submitted 2017-08-01; First posted 2017-08-03 (Actual); Results first posted 2021-06-04 (Actual); Last update posted 2021-06-04 (Actual); Status verified 2021-03

CONDITIONS: Diabetic Retinopathy
MeSH Terms: conditions — Diabetic Retinopathy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- BI 1467335 (Experimental)
  Interventions: Drug: BI 1467335
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BI 1467335 — Once daily
  Arms: BI 1467335
Drug: Placebo — Once daily
  Arms: Placebo

SUMMARY:
The main objective is to evaluate ocular and systemic safety and tolerability of BI 1467335 as well as whether BI 1467335 monotherapy has a potential to improve retinal lesions in patients with moderately severe Non-proliferative diabetic retinopathy (NPDR) (DRSS level 47) or severe Non-proliferative diabetic retinopathy (NPDR) (DRSS level 53), without Center-involved diabetic macular edema (CI-DME)

ELIGIBILITY:
Inclusion Criteria:

* Of legal age (according to local legislation, usually ≥ 18 years) at screening
* Male or female patients. Women of childbearing potential (WOCBP) must be ready and able to use two methods of contraception with at least one of them being a highly effective method of birth control per ICH M3 (R2) that result in a low failure rate of less than 1% per year when used consistently and correctly. A list of contraception methods meeting these criteria is provided in the patient information.
* Diagnosis of diabetes mellitus (type 1 or type 2):

  --Documented diabetes by American Diabetes Association (ADA) and/or World Health Organization criteria
* Glycosylated hemoglobin (HbA1c) ≤ 12% at screening
* Non-proliferative diabetic retinopathy (NPDR) without center-involved diabetic macular edema (CI-DME) in the study eye at screening with NPDR level 47 or level 53, as determined by the Central reading center (CRC) by using the DR severity scale (DRSS)
* Best corrected visual acuity ETDRS letter score ≥ 70 letters in the study eye at screening
* Media clarity, pupillary dilation and individual cooperation sufficient for adequate retinal examination including fundus photographs and Optical Coherence Tomography (OCT)
* Signed and dated written informed consent in accordance with ICH-GCP and local legislation prior to admission to the trial

Exclusion Criteria:

* Cataract surgery performed within 6 months prior to screening or planned during the trial in the study eye; or any additional eye disease in the study eye that, in the opinion of the investigator,could compromise or alter visual acuity during the course of the study (e.g. vein occlusion, uncontrolled intraocular pressure (IOP) >24 mmHg on optimal medical treatment, glaucoma with visual field loss, uveitis or other ocular inflammatory disease,vitreomacular traction, monocular vision, history of ischemic optic neuropathy, or genetic disorders such as retinitis pigmentosa)
* Active center-involved DME (CI-DME) on clinical examination and Optical Coherence Tomography (OCT) central subfield thickness in the study eye above 300 μm as measured by Optovue OCT or above 320 μm as measured by Heidelberg OCT
* Anterior segment and vitreous abnormalities in the study eye that would compromise the adequate assessment of the best corrected visual acuity or an adequate examination of the posterior pole
* Evidence of neovascularization on clinical examination including active neovascularization of the iris (small iris tufts are not an exclusion) or angle neovascularization in the study eye, ruled out by gonioscopy (documented in the last 4 weeks before screening or performed at screening)
* Prior pan-retinal photocoagulation (defined as ≥ 100 burns placed previously outside of the posterior pole) in the study eye
* Treatment of either DME or DR with macular laser within 3 months prior to screening, or intraocular injections of medication within 6 months prior to screening, and no more than 4 prior intraocular injections in the study eye at any time in the past
* Patients treated with Monoamine Oxidase (MAO) inhibitors or drugs that may have potential side effects due to MAO inhibition
* Current or planned, during the trial, use of medications known to be toxic to the retina, lens or optic nerve, or cause vision loss
* Patients who must or wish to continue the intake of other restricted medications or any drug considered likely to interfere with the safe conduct of the trial
* Estimated Glomerular filtration rate (eGFR) < 60 mL/min/1.73m2 calculated by Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation at screening, or where the investigator expects filtration rate is likely to drop below 60 mL/min/1.73m2 during the trial
* Alanine transaminase (ALT) or aspartate transaminase (AST) greater than 2.0-fold the upper limit of normal, or total bilirubin > 1.5x upper limit of normal.
* Uncontrolled arterial hypertension defined as a single measurement of systolic blood pressure >180 mmHg, or two consecutive measurements of systolic blood pressure > 160 mmHg and/or diastolic blood pressure >100 mmHg on optimal medical regimen at screening. If blood pressure is brought to ≤ 160/100 mmHg by antihypertensive treatment until randomization, individual can become eligible.
* Wolff-Parkinson-White Syndrome, baseline QTc > 450 ms (Fridericia's formula), family history of long QT, or on medication prolonging QT time at screening or planned initiation during the trial
* Diagnosis of a serious or unstable systemic or eye disease and other conditions that, in the clinical judgment of the investigator, are likely to interfere with the analyses of safety and efficacy in this study. Patients with an expected life expectancy of less than 2 years are also excluded.
* Active known or suspected chronic or relevant acute infections, such as HIV (Human Immunodeficiency Virus)\viral hepatitis, or tuberculosis. QuantiFERON® TB test and HBs Ag test will be performed during screening. Patients with a positive test result may participate in the study if further work up (according to local practice/guidelines) establishes conclusively that the patient has no evidence of active infection.
* Any documented active or suspected malignancy or history of malignancy within 5 years prior to screening, except appropriately treated basal cell carcinoma of the skin or in situ carcinoma of uterine cervix.
* Chronic alcohol or drug abuse or any condition that, in the investigator's opinion, makes them an unreliable study participant or unlikely to complete the trial
* Known hypersensitivity to any component of the trial drug and/or allergy to fluorescein dye
* Major surgery (major according to the investigator's assessment) performed within 12 weeks prior to randomization or planned during the trial, e.g. hip replacement
* Currently enrolled in another investigational drug trial, or less than 30 days or 5 times half-life of the investigational drug, whichever is longer, since ending another investigational drug trial from the screening visit in this trial or receiving other investigational treatment(s); patients participating in a purely observational trial will not be excluded.
* Previous randomization in this trial
* Women who are pregnant, nursing, or who plan to become pregnant while in the trial
* Any other clinical condition that, in the opinion of the investigator, would jeopardize patient safety while participating in this clinical trial.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2017-09-19 (Actual); Primary Completion 2020-05-14 (Actual); Study Completion 2020-05-14 (Actual)

CONTACTS AND LOCATIONS:
Locations (35):
- United States (16):
  - Trinity Research, Dothan, Alabama
  - Retinal Research Institute, LLC, Phoenix, Arizona
  - Retina-Vitreous Associates Medical Group, Beverly Hills, California
  - Stanford University Medical Center, Palo Alto, California
  - Florida Retina Institute, Orlando, Florida
  - Northwestern Medical Group, Chicago, Illinois
  - Raj K. Maturi, MD PC, Indianapolis, Indiana
  - Cumberland Valley Retina Consultants, PC., Hagerstown, Maryland
  - NJRetina, Teaneck, New Jersey
  - New York Eye and Ear Infirmary of Mount Sinai, New York, New York
  - Charlotte Eye Ear Nose and Throat Associates, PA, Charlotte, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Retina Research Institute of Texas, Abilene, Texas
  - Retina Research Center, PLLC, Austin, Texas
  - Retina Consultants of Houston, PA, Houston, Texas
- LKH-Univ. Hospital Graz, Graz, Austria
- Interbalkan Medical Center of Thessaloniki, Thessaloniki, Greece
- Italy (2):
  - Fondazione Centro San Raffaele del Monte Tabor, Milan
  - IRCCS Fondazione Bietti, Roma
- Oslo Universitetssykehus HF, Ullevål sykehus, Oslo, Norway
- Portugal (3):
  - CHUC - Centro Hospitalar e Universitário de Coimbra, EPE, Coimbra
  - Espaço Médico de Coimbra, Coimbra
  - CHULC, EPE - Hospital Sto. António Capuchos, Lisbon
- Spain (4):
  - Hospital Dos de Maig, Barcelona
  - Hospital Vall d'Hebron, Barcelona
  - Hospital Clínico San Carlos, Madrid
  - Hospital Miguel Servet, Zaragoza
- United Kingdom (7):
  - Bradford Royal Infirmary, Bradford
  - Bristol Eye Hospital, Bristol
  - Frimley Park Hospital, Frimley
  - Moorfields Eye Hospital, London
  - Royal Victoria Infirmary, Newcastle upon Tyne
  - Hospital of St Cross, Rugby
  - Sunderland Eye Infirmary, Sunderland

REFERENCES:
- See also: Related Info — https://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A study evaluated safety and tolerability of 12-week treatment of oral BI 1467335 compared to placebo in patients with moderately severe to severe non-proliferative diabetic retinopathy without center-involved diabetic macular edema and explored the efficacy of BI 1467335 on improvement of diabetic retinopathy.
Pre-assignment Details: All subjects were screened for eligibility prior to participation in the trial. Subjects attended a specialist site which ensured that they (the subjects) strictly met all inclusion and none of the exclusion criteria.
  Subjects were not to be allocated to a treatment group if any of the entry criteria were violated.
Groups:
- BI 1467335 10 mg: 2 film coated tablets of 5 milligram (mg) BI 1467335 (Total: 10 mg) were taken orally once daily for a treatment period of 12 weeks with 12 weeks of follow-up.
- Placebo: 2 film coated tablets of matching placebo were taken orally once daily for a treatment period of 12 weeks with 12 weeks of follow-up.
Period: Overall Study
Arm/Group | BI 1467335 10 mg | Placebo
Started | 40 | 39
Completed | 35 | 37
Not Completed | 5 | 2
Not completed — Prohibited medication given due to hospital stay | 1 | 0
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Protocol Violation | 1 | 1
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Population: Treated set (TS): the TS consists of all patients who were treated with at least one dose of trial drug (BI 1467335 or placebo).
Groups:
- Total: Total of all reporting groups
Arm/Group | BI 1467335 10 mg | Placebo | Total
Number analyzed (Participants) | 40 | 39 | 79
Age, Continuous [Mean (Standard Deviation); unit: Years] | 52.5 (10.8) | 53.1 (13.3) | 52.8 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 14 | 28
  Male | 26 | 25 | 51
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 18 | 15 | 33
  Not Hispanic or Latino | 22 | 24 | 46
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 1 | 4 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 3 | 6
  White | 36 | 31 | 67
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Any Ocular Adverse Events Over the On-treatment Period
Description: Percentage of participants with any ocular adverse events over the on-treatment period was reported.
Time Frame: On-treatment period: from first dose of study drug until end of follow-up period, up to 24 weeks.
Population: as for baseline characteristics
Measure: Number; unit: Percentage of participants
Arm/Group | BI 1467335 10 mg | Placebo
Number analyzed (Participants) | 40 | 39
Percentage of participants | 35.0 | 23.1

2. Secondary Outcome: Percentage of Participants With at Least 2 Steps Improvement From Baseline in the Study Eye on the Diabetic Retinopathy Severity Scale (DRSS) at Week 12
Description: 7-field or modified 4-field digital fundus photographs was obtained from both eyes by a qualified person according to the imaging manual to collect all data for the assessment of the Early Treatment Diabetic Retinopathy Study (ETDRS) Diabetic Retinopathy Severity Scale (DRSS). The images was sent to the independent central reading center who performs the grading on the basis of the DRSS. The DRSS ranges from level 10 (Diabetic retinopathy absent) to level 85 (advanced proliferative Diabetic retinopathy).
Time Frame: At baseline and at Week 12.
Population: Full analysis set (FAS): the FAS consists of all the patients who were randomized, treated with at least one dose of BI 1467335/placebo and have baseline and one on-treatment Diabetic Retinopathy Severity Scale assessment. Only patients with non-missing endpoint results were included in the analysis.
Measure: Number; unit: Percentage of participants
Arm/Group | BI 1467335 10 mg | Placebo
Number analyzed (Participants) | 35 | 34
Percentage of participants | 5.7 | 0.0
Statistical Analysis 1: Comparison: BI 1467335 10 mg vs Placebo; Test type: Other; Chan and Zhang method; 95% confidence interval was calculating using the Chan and Zhang method; Risk Difference (RD) = 0.057, 95% CI 2-sided [-0.053 to 0.192], Standard Error of Mean 0.039 — Risk difference of BI 1467335 10 milligram (mg) group minus Placebo group

3. Secondary Outcome: Percentage of Participants With Adverse Events Other Than Ocular Adverse Events Over On-treatment Period
Description: Percentage of participants with adverse events other than ocular adverse events over on-treatment period was reported.
Time Frame: On-treatment period: from first dose of study drug until end of follow-up period, up to 24 weeks.
Population: as for baseline characteristics
Measure: Number; unit: Percentage of participants
Arm/Group | BI 1467335 10 mg | Placebo
Number analyzed (Participants) | 40 | 39
Percentage of participants | 55.0 | 82.1

ADVERSE EVENTS:
Time Frame: From first dose of study drug until end of follow-up period, up to 24 weeks.
Description: Treated set (TS): the TS consists of all patients who were treated with at least one dose of trial drug (BI 1467335 or placebo).
Arm/Group | BI 1467335 10 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/39
Serious Adverse Events (participants affected / at risk) | 7/40 | 4/39
Other Adverse Events (participants affected / at risk) | 16/40 | 25/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BI 1467335 10 mg (N=40) | Placebo (N=39)
Angina pectoris (Cardiac disorders) | 1 | 0
Visual acuity reduced (Eye disorders) | 1 | 0
Impaired gastric emptying (Gastrointestinal disorders) | 1 | 0
Pancreatitis chronic (Gastrointestinal disorders) | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0
Cellulitis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0
Liver function test increased (Investigations) | 1 | 0
Cervix carcinoma stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Dysarthria (Nervous system disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BI 1467335 10 mg (N=40) | Placebo (N=39)
Diabetic retinopathy (Eye disorders) | 3 | 2
Abdominal pain upper (Gastrointestinal disorders) | 2 | 2
Diarrhoea (Gastrointestinal disorders) | 0 | 3
Nausea (Gastrointestinal disorders) | 2 | 6
Vomiting (Gastrointestinal disorders) | 0 | 2
Localised infection (Infections and infestations) | 0 | 2
Nasopharyngitis (Infections and infestations) | 2 | 5
Urinary tract infection (Infections and infestations) | 1 | 2
Alanine aminotransferase increased (Investigations) | 0 | 2
Blood glucose increased (Investigations) | 1 | 3
Gamma-glutamyltransferase increased (Investigations) | 0 | 2
Glucose urine present (Investigations) | 1 | 2
Lipase increased (Investigations) | 0 | 2
Protein urine present (Investigations) | 0 | 3
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 2
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 2
Headache (Nervous system disorders) | 7 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results.

Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days.

BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2019-04-11): https://cdn.clinicaltrials.gov/large-docs/63/NCT03238963/Prot_000.pdf
  • Statistical Analysis Plan (2020-06-29): https://cdn.clinicaltrials.gov/large-docs/63/NCT03238963/SAP_001.pdf